CLINICAL TRIAL: NCT03993587
Title: The Effect of Head and Shoulder Positioning on the Cross-sectional Area and Location of the Subclavian Vein in Obese Adults
Brief Title: The Effect of Head and Shoulder Positioning on the Cross-sectional Area of the Subclavian Vein in Obese Adults
Status: Completed | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: P2019-192
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Normal Volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound assessment of vessels — Subclavian vein and related structures are examined using ultrasonography

SUMMARY:
In the present study, the cross-sectional area of subclavian vein, and the depth of the SCV from the skin are assessed in different head positions (neutral, rotation to ipsilateral or contralateral sides) and different shoulder positions (neutral or lowered) in spontaneous breathing obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy obese adults (BMI ≥ 30)

Exclusion Criteria:

* Medication affecting vascular elasticity History of central venous catheterization or clavicle fracture History of lung surgery, operation of chest cage

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy obese adults (BMI ≥ 30)
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cross-sectional area of subclavian vein | through the completion of assessment, an average of 1 hr
  Cross-sectional area of subclavian vein is assessed.

SECONDARY OUTCOMES:
Depth of subclavian vein from skin | through the completion of assessment, an average of 1 hr
  Depth of subclavian vein from skin is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No